CLINICAL TRIAL: NCT03565523
Title: The Effect of Dietary Nitrate Supplementation on Linear Running Sprint Performance, Agility and Vertical Jump Performance in a Rested and Fatigued State
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PEP-1607
Record Dates: First submitted 2018-06-06; First posted 2018-06-21 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Exercise Performance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Beet shot (Experimental): Containing 385 mg nitrate
  Interventions: Other: Beetroot
- Placebo beverage (Placebo Comparator): <0.1 mmol nitrate in sucrose solution with beet coloring
  Interventions: Other: Placebo beverage

INTERVENTIONS:
Other: Beetroot — Containing 385 mg nitrate
  Arms: Test Beet shot
Other: Placebo beverage — <0.1 mmol nitrate in sucrose solution with beet coloring
  Arms: Placebo beverage

SUMMARY:
Dietary nitrate (NO3-) supplementation has been shown to improve skeletal muscle contractility and fatigue resistance, particularly in fast-twitch (type II) muscle fibers. Furthermore, NO3- supplementation has been shown to speed reaction time. Taken together, these findings suggest that NO3- ingestion may be ergogenic during all-out sprint running and reactive agility tasks. Moreover, increasing muscle force production at high contraction speeds would be expected to translate into improved muscle power and, subsequently, improved performance in very explosive forms of exercise, such as vertical jumping. Therefore, the purpose of this investigation is to assess the effect of short term (5 days) NO3- supplementation on linear running sprint performance, reactive agility and vertical jump performance in a rested and fatigued state.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants in self-reported good general health as assessed by the standard procedures described below and specifically meeting normal blood pressure range (systolic: 100-135, diastolic: 60-90) and body mass index (BMI) range (16.0-29.9)
2. Range of 18-45 years of age
3. Participants must participate in an intermittent exercise based sport (e.g. soccer, rugby, hockey), at a competitive level (i.e. competes in officiated matches/games).
4. Understanding of the procedures to be undertaken as part of the study
5. Willingness to participate in exercise testing and follow supplementation guidelines and other instructions provided by the experimenter
6. Informed, voluntary, written consent to participate in the study

Exclusion Criteria:

1. Known pulmonary, cardiovascular or metabolic disease
2. Food allergies including phenylketonurea (PKU)
3. Current regular use of any dietary supplement (excluding macronutrient based supplements) or previous use of any dietary supplement in the past 6 months that is known to have a lasting effect.
4. Blood donation within 3 months prior to the start of the study
5. Substance abuse within 2 years of the start of the study
6. Smoking
7. Any prescription and non-prescription medication which may impact saliva production (antidepressants, diuretics, analgesics, antihistamines, anti-hyper/hypo-tensives, anti-anxiety, appetite suppressants).
8. Current or previous use of phosphodiesterase 5 (PDE5) inhibitors.
9. Participation in another clinical trial within past 4 weeks.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Linear running sprint time | 5 days
  Linear running sprint in a rested and fatigued state

CONTACTS AND LOCATIONS:
Overall Officials: Andy Jones, PhD, Principal Investigator — University of Exeter, Sport and Health Sciences department

IPD SHARING:
Plan to Share IPD: No